CLINICAL TRIAL: NCT06898541
Title: Impact of the Coronary Sinus Reducer on Coronary Flow Reserve and Symptoms in Patients With Coronary Microvascular Disease
Brief Title: Coronary Sinus Reducer in Coronary Microvascular Disease
Acronym: REDUCE CMD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Radboud University Medical Center (Other); Maasstad Hospital, Rotterdam (Unknown); VieCuri, Venlo, the Netherlands (Unknown)
Responsible Party: Principal Investigator, Tim P. van de Hoef, Principal Investigator, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REDUCE CMD
Record Dates: First submitted 2025-01-04; First posted 2025-03-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Angina (Stable); Coronary Microvascular Disease
Keywords: Angina; Coronary microvascular disease; Coronary sinus reducer
MeSH Terms: conditions — Angina, Stable; Microvascular Angina; Angina Pectoris | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham (Sham Comparator): Patients in this arm undergo a sham CSR procedure.
  Interventions: Other: Sham CSR procedure
- CSR arm (Experimental): Patients in this arm undergo coronary sinus reducer implantation.
  Interventions: Device: Coronary sinus reducer

INTERVENTIONS:
Device: Coronary sinus reducer — Implantation of a Coronary Sinus Reducer device
  Other Names: reducer
  Arms: CSR arm
Other: Sham CSR procedure — Patients will undergo a complete sham CSR implantation procedure without actual deployment of the CSR.
  Other Names: Sham
  Arms: Sham

SUMMARY:
Coronary microvascular dysfunction (CMD) is a common cause of treatment- resistant angina that lacks evidence-based treatment options. The coronary sinus reducer (CSR) is an hourglass-shaped stainless steel mesh, designed to create a controlled narrowing of the coronary sinus (CS). By augmenting CS pressure, CSR implantation was shown to improve myocardial perfusion, potentially providing a novel treatment for patients with CMD. REDUCE CMD is a placebo-controlled study of CSR in 50 patients with CMD. The main study endpoints are the change in coronary flow reserve from baseline to 6 months in the CSR-arm versus the placebo arm, and the difference in number of daily episodes of angina recorded on the ORBITA-app at 6 month follow-up in the CSR-arm versus the placebo arm.

ELIGIBILITY:
Inclusion criteria

1. Coronary microvascular dysfunction in the left anterior descending coronary artery (LAD) as expressed by abnormal absolute coronary flow reserve (CFR<2.5) confirmed during the index study procedure using the continuous thermodilution technique and saline-induced coronary hyperaemia.
2. Angina - Canadian Cardiovascular Society Class II-IV on at least two anti-anginals or maximally tolerated medical therapy if less than two.
3. Patient understands the nature of the procedure and provides written informed consent for the study prior to enrolment.

Exclusion criteria

1. Age < 18 years.
2. Absence of symptoms reported on the ORBITA-app during the 2-week screening period.
3. Presence of hemodynamically significant epicardial stenoses based on both non- hyperaemic pressure ratio (NHPR; iFR≤0.89, or RFR≤0.89, or dFR/dPR≤0.89) or fractional flow reserve (FFR≤0.80) assessments.
4. Prior positive acetylcholine provocation test with respect to epicardial vasospasm following the COVADIS criteria.
5. Mean right atrial pressure ≥15 mmHg
6. Severe pulmonary hypertension.
7. Coronary sinus anatomy not suitable for CSR implantation.
8. Pregnancy or planned pregnancy within the next 12 months.
9. Recent acute coronary syndrome (within 3 months).
10. Recent revascularization with PCI (within 6 months).
11. Severe arrhythmias, including chronic atrial fibrillation with persistent rapid ventricular response (>100bpm despite medication).
12. Indication for cardiac resynchronization therapy.
13. Severe left ventricular impairment (left ventricular ejection fraction <35%).
14. NYHA class IV or decompensated heart failure or hospitalization due to heart failure within 90 days before the index procedure.
15. Recent implantation of a permanent pacemaker or defibrillator lead in the right ventricle or atrium (within 90 days before the index procedure).
16. Presence of a pacemaker lead in the coronary sinus.
17. Severe valvular heart disease.
18. History of tricuspid valve replacement or repair.
19. Contra-indication to short term dual antiplatelet therapy or lifelong aspirin treatment.
20. Currently enrolled in another investigational device or drug trial that has not completed the primary endpoint or that clinically interferes with the current study endpoints.
21. Known inability to tolerate contrast medium.
22. Life expectancy <1 year.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-20 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in coronary flow reserve | 6 months
  Change in coronary flow reserve from baseline to 6 months in the CSR-arm versus the placebo arm (measured by the continuous flow thermodilution technique using saline-induced coronary hyperaemia).
Angina episodes | 6 months
  Difference in number of daily episodes of angina recorded on the ORBITA-app at 6 month follow-up in the CSR-arm versus the placebo arm.

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Maasstad Ziekenhuis, Rotterdam
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No